CLINICAL TRIAL: NCT00194402
Title: SLIM: Combined Effects of Slo-Niacin and Atorvastatin on Lipoproteins and Inflammatory Markers
Brief Title: SLIM: Combined Effects of Slo-Niacin and Atorvastatin on Lipoproteins and Inflammatory Markers in Hyperlipidemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Upsher-Smith Laboratories (Industry)
Responsible Party: Robert H. Knopp, MD, Professor of Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03-6262-A
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2008-08-21 (Estimated); Status verified 2008-08

CONDITIONS: Dyslipidemia
Keywords: cholesterol; dyslipidemia; hypercholesterolemia; C-reactive protein
MeSH Terms: conditions — Dyslipidemias; Hypercholesterolemia | interventions — Niacin; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Atorvastatin 10 mg for 12 weeks followed by Slo-Niacin (titrated from 500 to 1500 mg over 8 weeks) taken with atorvastatin 10 mg for an additional 12 weeks
  Interventions: Drug: Slo-Niacin, atorvastatin
- 2 (Active Comparator): Slo-Niacin (titrated from 500 to 1500 mg over 8 weeks) for 12 weeks followed by atorvastatin 10 mg taken with Slo-Niacin 1500 mg for an additional 12 weeks
  Interventions: Drug: Slo-Niacin, atorvastatin

INTERVENTIONS:
Drug: Slo-Niacin, atorvastatin — Atorvastatin 10 mg qd for 12 or 24 weeks. Time-released niacin 1500 mg qd (titrated from 500mg to 1000mg and then to 1500 mg at 4 week intervals) taken for 12 or 24 weeks.
  Other Names: Lipitor (R) (Atorvastatin); Slo-Niacin (R) (time-release niacin

SUMMARY:
Slo-Niacin and atorvastatin (Lipitor) are both drugs that lower cholesterol. In this research, we will compare the effectiveness of Slo-Niacin and atorvastatin taken alone and together. This study will help show how the individual benefits of the two drugs taken separately can be combined when taken together.

DETAILED DESCRIPTION:
Combined niacin and a statin treatment has greater potential value than either agent alone for the dyslipidemia of insulin resistance, obesity and the metabolic syndrome. The efficacy of Slo-Niacin and atorvastatin has not been formally examined in this setting.

Methods: Forty-four dyslipidemic men and women (LDL-C >130mg/dL and below average HDL-C (<55 in women and <45 in men) were randomized to a 3 month course of atorvastatin 10 mg or Slo-Niacin increased monthly at doses of 500, 1000 and 1500 mg/day. The alternate drug was added in the second 3-month segment. Lipid profiles and transaminase measurements were obtained monthly and full lipoprotein quantifications, apoproteins, remnant like lipoproteins (RLP), LDL buoyancy, glucose, insulin, and C-reactive protein were measured at the end of each 3-month sequence. Results: Mean entry lipids were (mg/dL) TG 187, LDL-C 171, HDL-C 39. Mean BMI was 32.6 Kg/M2. When Slo-Niacin and atorvastatin were given alone, respective decreases in triglyceride (TG) were 18% and 10%, LDL-C 12% and 36% and non-HDL-C 15% and 36%. HDL-C increased 8% and 6%, respectively. Combined therapy decreased median TG 33% and mean LDL-C 43% and increased mean HDL-C 10%. Mean hs CRP decreased 23% and RLP 44.5% in the combined groups. Conclusions: Slo-Niacin with atorvastatin improves all lipoprotein fractions, RLP and hsCRP in combined hyperlipidemia. The reduction of LDL with the drug combination is equivalent to that obtained with 20-80 mg of atorvastatin alone.

ELIGIBILITY:
Inclusion Criteria:

* LDL-C > 130 mg/dL
* HDL-C <= 45 mg/dL in men and <= 55 mg/dL in women

Exclusion Criteria:

* history of hypersensitivity to any statin, niacin or aspirin
* diagnosis of diabetes or a fasting glucose > 125 mg/dL
* hyper or hypothyroidism (unless treatment stable)
* meet other health, medication, and logistical criteria

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2003-08; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
LDL-C change for atorvastatin 10 mg, Slo-Niacin 1500 mg, and the two together. | Change from baseline to 12 weeks and end of intervention

SECONDARY OUTCOMES:
Change in HDL-C, HDL2-C, HDL3-C, LDL-C:HDL-C, triglyceride, remnant lipoprotein, apoproteins A-I and B, LDL buoyancy, hsCRP, glucose, insulin, and SGOT. | Change from baseline to end of 12 weeks and/or end of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Robert H. Knopp, MD, Principal Investigator — Northwest Lipid Research Clinic, University of Washington
Locations (1):
- Northwest Lipid Research Clinic, University of Washington, Seattle, Washington, United States